CLINICAL TRIAL: NCT03053232
Title: Purse String Suture Device Versus Endoclip in the Treatment of Immediate Endoscopic Procedure Associated Gastrointestinal Perforation
Brief Title: Purse String Suture Device vs. Endoclip for Immediate Endoscopic Procedure Associated Gastrointestinal Perforation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307-LM
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Intervention; Gastrointestinal Perforation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purse string suture device (Experimental): Use of purse string suture device to close gastrointestinal perforation.
  Interventions: Device: Purse string suture device
- Endoclips (Active Comparator): Use of endoclips to close gastrointestinal perforation.
  Interventions: Device: Endoclips

INTERVENTIONS:
Device: Purse string suture device — Using purse string suture device to close gastrointestinal perforation under endoscopy.
  Arms: Purse string suture device
Device: Endoclips — Using endoclips to close gastrointestinal perforation under endoscopy.
  Arms: Endoclips

SUMMARY:
Nowadays, endoscopic techniques have been applied for diagnosing and treating a variety of gastrointestinal diseases, such as endoscopic submucosal dissection (ESD) and endoscopic mucosal resection (EMR)technique for removing early gastrointestinal mucosal cancers. Endoscopic procedure associated gastrointestinal perforation is one of the the most severe complications, which is associated with high morality and needs timely detection and effective treatment in clinical practice.Over 90% procedure associated gastrointestinal perforation occurs immediately within 24 h after endoscopic procedure.Endoclips have been widely used in closing the immediate gastrointestinal perforations, but the location of the endoclips could influence the effective rate, limiting its application. In addition, multiple endoclips should be placed under endoscopy for a relatively large perforation, which could increase the medical cost and the procedure time. At recent, a new purse string suture device (LeoMed, China) has been developed by us and introduced to the clinicalmanagement of such patients with procedure associated gastrointestinal perforations. Clinical data validated that the usage of this new purse string suture in treating immediate procedure associated perforations was greatly convenient and effective with very low reoperation rate and postoperative complication rate. A specially designed loop was equipped in this device, which could be tightened under endoscopy. Thus, compared with the placement of endoclips, this device could be more convenient and effective in completely closing the gastrointestinal perforations.This study will test whether purse string suture device will increase the effectiveness of closingimmediate procedure associated gastrointestinal perforationsunder endoscopyin a randomized controlled trialby comparing the use of purse string suture deviceand endoclips.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing the use of purse string suture device versus endoclips for closing procedure associated gastrointestinal perforation under endoscopy, which is one of the most severe complications and needs timely treatment. Endoclips have been widely used in closing the gastrointestinal perforations, but the location of the endoclips could significantly influence the effective rate. In addition, multiple endoclips will be needed for a relatively large perforation, which could increase the medical cost and the procedure time. At recent, a new purse string suture device has been developed and introduced to the clinicalmanagement of such patients with gastrointestinal perforations. A loop was equipped in this device, which could be tightened. Thus, compared with endoclips, this device could be more convenient and effective in completely closing the gastrointestinal perforations. This study will test whether purse string suture device will increase the effectiveness of treating procedure associated gastrointestinal perforations under endoscopy in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 Years
* Immediate procedure associated gastrointestinal perforation (i.e. post-ESD perforation, post-EMR perforation；complications of endoscopic examination and procedure)
* American Society of Anesthesiology risk class 1, 2 or 3

Exclusion Criteria:

* Patients <18 years
* Patients with thrombocytopenia (platelet count < 50,000/microL) or elevated - International Normalized Ratio (INR > 1.5)
* Hemodynamic instability
* Pregnancy and lactation
* Patients who are unable or unwilling to give an informed consent
* Chronic fistula following abdominal surgery
* Pyriform fossa perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Technique success rate | 1 year
  Percentage of patients who successfully receive endoscopical interventions

SECONDARY OUTCOMES:
Effective rate | 1 year
  Percentage of patients whose clinical symptoms are alleviated and perforations closed
Postoperative complication rate | 1 year
  Percentage of patients who have complications including death after procedure
Reoperation rate | 1 year
  Percentage of patients who need a secondary operation
Operation time | 1 year
  The time length of the endoscopic operation will be recorded in the unit of minute.
Postoperative pain | 1 year
  Postoperative pain will be evaluated on a visula analogue score (VAS).
Postoperative hospitalization | 1 year
  The length of the hospitalizatioin after operation will be recorded in the unit of day.
Time to resume diet | 1 year
  When the patients resume diet will be monitored and recorded.
Medical cost | 1 year
  The medical cost for the operation and hospitalization will be recorded and collected.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schultz JK, Yaqub S, Wallon C, Blecic L, Forsmo HM, Folkesson J, Buchwald P, Korner H, Dahl FA, Oresland T; SCANDIV Study Group. Laparoscopic Lavage vs Primary Resection for Acute Perforated Diverticulitis: The SCANDIV Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1364-75. doi: 10.1001/jama.2015.12076. PMID 26441181
- [Background] Tan S, Wu G, Zhuang Q, Xi Q, Meng Q, Jiang Y, Han Y, Yu C, Yu Z, Li N. Laparoscopic versus open repair for perforated peptic ulcer: A meta analysis of randomized controlled trials. Int J Surg. 2016 Sep;33 Pt A:124-32. doi: 10.1016/j.ijsu.2016.07.077. Epub 2016 Aug 5. PMID 27504848